CLINICAL TRIAL: NCT04547010
Title: Effects of Soy Isoflavone on Bone Health Among Saudi Female Students Imam Abdulrahman Bin Faisal University.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Tunny Sebastian, Assistant Professor, Imam Abdulrahman Bin Faisal University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-UGS-2018-03-273
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Soy Isoflavone Effect; Bone Density, Low; Bone Density Increased
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteosclerosis

STUDY DESIGN:
Intervention Model Description: Pre-post Quasi experimental study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): In four weeks of intervention study the participants instructed to receive (60 mg) of soy-isoflavone supplement per day, after this period the Bone Mineral Density was assessed by Dual X-ray Absorptiometry scan to evaluate the effect of soy-isoflavone supplement on Bone mineral density.
  Interventions: Dietary Supplement: Soy Isoflavone supplement

INTERVENTIONS:
Dietary Supplement: Soy Isoflavone supplement — Participants received 60 mg of soy-isoflavone supplement per day.

SUMMARY:
Low bone mineral density (BMD) has recently increased among young women. Soy Isoflavone as a food supplement, has been found to have potent effect on bone health in postmenopausal women. However, the effect of soy isoflavone on pre-menopausal is not well understood. This research is done to examine the effect of soy isoflavones on BMD among young university female students.

ELIGIBILITY:
Inclusion Criteria:

* female
* University students
* aged between 18-25 years

Exclusion Criteria:

* Study participants who use medications and suffer from diseases that may interfere or effect on BMD, use calcium and vitamin D supplements and who suffer from glucose 6 phosphate deficiency (G6PD) were excluded from the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No